CLINICAL TRIAL: NCT01653912
Title: An Open-Label Phase I/II Study of GSK2110183 in Combination With Carboplatin and Paclitaxel in Subjects With Platinum-Resistant Ovarian Cancer
Brief Title: Dose-finding Study in Platinum-Resistant Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Accenture (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKB116611; 2012-002483-27 (EudraCT Number)
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2017-08

CONDITIONS: Recurrent Platinum-resistant Ovarian Cancer
Keywords: cancer; ovarian; platinum-resistant
MeSH Terms: conditions — Neoplasms | interventions — GSK2110183; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK2110183, carboplatin and paclitaxel (Experimental): Subjects will be treated with a maximum of six doses of carboplatin + paclitaxel in combination with continuous daily GSK2110183 followed by single agent GSK2110183 at the single-agent MTD of 125 mg or above oral daily.
  Interventions: Drug: GSK2110183 in combination with carboplatin and paclitaxel

INTERVENTIONS:
Drug: GSK2110183 in combination with carboplatin and paclitaxel — Phase I is a dose escalation evaluation of increasing doses of GSK2110183 administered on a continuous daily schedule in combination with carboplatin AUC 5 and paclitaxel 175mg/m2 given every three weeks for a maximum 6 cycles. The dosing regimen identified in Phase I will then be evaluated in Phase II, a single arm study focused on clinical efficacy. Treatment with the three drug regimen will continue for a maximum of 6 x 21 day cycles followed by continuous GSK2110183 at the single agent MTD. Subjects may continue on study drug until progression, death or unacceptable toxicity.
  Other Names: Taxol (paclitaxel); Paraplatin (carboplatin); AKT Inhibitor

SUMMARY:
* Dose-finding study of GSK2110183 administered in combination with carboplatin and paclitaxel to any subject with recurrent ovarian cancer.
* Safety and efficacy study of GSK2110183 administered in combination with carboplatin and paclitaxel to subjects with platinum-resistant ovarian cancer.

DETAILED DESCRIPTION:
PKB116611 is an open-label Phase I/II study of the investigational drug GSK2110183 given in combination with carboplatin and paclitaxel to subjects with recurrent ovarian cancer. Phase I is a dose escalation evaluation of daily oral doses of GSK2110183 administered in combination with every 3 week carboplatin and paclitaxel to any subject with recurrent ovarian cancer. Phase II is a single arm evaluation of the clinical efficacy of the combination identified in Phase I to subjects with platinum-resistant ovarian cancer.

ELIGIBILITY:
Phase I Inclusion Criteria:

* Female, 18 years of age as of signing the informed consent form, capable of giving/complying with written informed consent
* Histologically or cytologically confirmed serous ovarian cancer (includes primary peritoneal and Fallopian tube)
* Negative serum pregnancy test in women of childbearing potential within 14 days of first dose of treatment, agree to use effective contraception during/after (6 months post dose of paclitaxel or 30 days post dose GSK2110183 whichever is longer)
* Performance Status score of 0-2 according to the ECOG scale.
* Able to swallow and retain oral medication
* Subjects diagnosed previously with Type 2 diabetes must have been diagnosed ≥ 6 months prior to enrollment
* Prior treatment-related toxicities (except for alopecia) must be ≤ Grade 1 according to NCI-CTCAE (Version 4.0 [NCI, 2009]) at the time of treatment allocation OR ≤ Grade 2 and stable for 4 weeks or longer at the time of screening evaluation. Exception: Subjects with peripheral neuropathy >/= Grade 2 will NOT be eligible
* Adequate organ system function

Phase II Inclusion Criteria:

Cohort A

* Phase I criteria
* Documented complete or partial response by RECIST to at least 1 prior platinum-based therapy
* Progression defined by either (1) RECIST v1.1 criteria or (2) GCIG CA 125 criteria associated with symptoms necessitating treatment between 1 and 6 months of prior platinum-based therapy either in adjuvant or metastatic setting
* Subjects allowed to have a maximum of one non-platinum-based therapy between the onset of platinum resistance
* Must have radiologically measurable disease i.e. presenting with at least one measurable lesion per RECIST 1.1

Cohort B

* Phase I criteria
* Documented complete or partial response by RECIST to at least 1 prior platinum-based therapy
* Progression defined by either (1) RECIST v1.1 criteria or (2) GCIG CA 125 criteria associated with symptoms necessitating treatment while being treated with a regimen containing carboplatin and paclitaxel (or within 4 weeks of completing treatment)
* Subjects will be required to start on treatment within 8 weeks after the last infusion of chemotherapy and may not have had any other anti-cancer therapy in the intervening time
* Must have radiologically measurable disease i.e. presenting with at least one measurable lesion per RECIST 1.1
* Additional restrictions on number of prior therapies may be added to eligibility criteria based on emerging data

Exclusion Criteria:

* History of another malignancy (some exceptions may apply)
* Serious and/or unstable pre-existing medical or psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures
* Current use of prohibited medication during treatment.
* Chemotherapy, immunotherapy, or other anti-cancer therapy within 14 days prior to the first dose study drug
* Radiotherapy prior to initiation of therapy (some exceptions may apply)
* Contraindications (identified by the investigator) to the doses of carboplatin and/or paclitaxel
* History of reduction in standard of care paclitaxel dose for peripheral neuropathy
* No known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to drugs similar or related to GSK2110183
* No known delayed hypersensitivity reaction or idiosyncratic reaction to drugs similar to carboplatin or paclitaxel (some exceptions may apply)
* Prior use of a drug that targets AKT including perifosine
* History of Type 1 diabetes
* Gastrointestinal disease or other condition that could affect absorption or predispose subject to gastrointestinal ulceration
* Mucosal or internal bleeding
* Major surgery within the last four weeks
* Infection requiring parenteral or oral anti-infective treatment
* Severe or uncontrolled systemic diseases
* Brain metastases and/or leptomeningeal disease
* QTcF interval ≥ 470 msecs
* Bundle branch block, pacemaker or clinically significant ECG abnormalities including 2nd degree (Type II) or 3rd degree atrioventricular (AV) block
* History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty,stenting or bypass grafting within six months of Screening
* Class II, III or IV heart failure as defined by the NYHA functional classification system
* Pregnant or lactating female
* Malignancies related to HIV or solid organ transplant; history of known HIV, history of know HBV surface antigen positivity (subjects with documented laboratory evidence of HBV clearance may be enrolled) or positive HCV antibody

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-11; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Brigandi, MD, PhD, FAAP, Study Director — GlaxoSmithKline; Anne L Hamilton, Principal Investigator — Royal Women's Hospital; Sarah P Blagden, Principal Investigator — Imperial College Healthcare NHS Trust; Linda Mileshkin, Principal Investigator — Peter MacCallum Cancer Centre, Australia; Shirley S Wong, Principal Investigator — Western Hospital; Andrew Dean, Principal Investigator — Sir Charles Gairdner Hospital; Marcia Hall, Principal Investigator — Mount Vernon Cancer Center; Bhawana Awasthy, MD, Study Director — Syneos Health
Locations (10):
- Australia (5):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Western Hospital, Footscray, Victoria
  - Royal Women's Hospital, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Russia (2):
  - Medical Radiology Scientific Center of Ministry of Healthcare and Social Development of RF, Omskaya
  - City Clinical Oncology Dispensary, Saint Petersburg
- United Kingdom (3):
  - Mount Vernon Cancer Center, Northwood, Middlesex, London
  - Royal Surrey County Hospital NHS Foundation Trust, Guildford, Surry
  - Imperial College Healthcare NHS Trust, London

REFERENCES:
- [Derived] Blagden SP, Hamilton AL, Mileshkin L, Wong S, Michael A, Hall M, Goh JC, Lisyanskaya AS, DeSilvio M, Frangou E, Stronach EA, Gopalakrishna P, Meniawy TM, Gabra H. Phase IB Dose Escalation and Expansion Study of AKT Inhibitor Afuresertib with Carboplatin and Paclitaxel in Recurrent Platinum-resistant Ovarian Cancer. Clin Cancer Res. 2019 Mar 1;25(5):1472-1478. doi: 10.1158/1078-0432.CCR-18-2277. Epub 2018 Dec 18. PMID 30563934

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 10 centers in 3 countries (United Kingdom, Australia, and Russia)
Pre-assignment Details: As described in Statistical Analysis Plan (SAP) dated 14-Jul-2015, as there were <10 subjects in Cohort B (n=2), data was summarized in phase 2 total column but not presented in a separate column for Cohort B.
Groups:
- Phase 1 (Dose Escalation)-Cohort 1: GSK2110183 50 mg: GSK2110183 50 mg capsule by mouth daily in combination with carboplatin Area Under the Curve (AUC) 5 and paclitaxel 175 mg/m2 given intravenously every 3 weeks for a maximum 6 cycles.
- Phase 1 (Dose Escalation)-Cohort 1.5: GSK2110183 75 mg: GSK2110183 75 mg capsule by mouth daily in combination with carboplatin AUC 5 and paclitaxel 175 mg/m2 given intravenously every 3 weeks for a maximum 6 cycles.
- Phase 1 (Dose Escalation)-Cohort 2: GSK2110183 100 mg: GSK2110183 100 mg capsule by mouth daily in combination with carboplatin AUC 5 and paclitaxel 175 mg/m2 given intravenously every 3 weeks for a maximum 6 cycles.
- Phase 1 (Dose Escalation)-Cohort 3: GSK2110183 125 mg: GSK2110183 125 mg capsule by mouth daily in combination with carboplatin AUC 5 and paclitaxel 175 mg/m2 given intravenously every 3 weeks for a maximum 6 cycles.
- Phase 1 (Dose Escalation)-Cohort 4: GSK2110183 150 mg: GSK2110183 150 mg capsule by mouth daily in combination with carboplatin AUC 5 and paclitaxel 175 mg/m2 given intravenously every 3 weeks for a maximum 6 cycles.
- Phase 2 (Treatment Group): GSK2110183 125 mg (MTD): The dosing regimen identified in Phase I will then be evaluated in Phase II, a single arm study focused on clinical efficacy. GSK2110183 125 mg (MTD) capsule by mouth daily in combination with carboplatin AUC 5 and paclitaxel 175 mg/m2 given intravenously every 3 weeks for a maximum 6 x 21 day cycles followed by continuous GSK2110183 150 mg capsule by mouth daily until progression, death or unacceptable toxicity.
Period: Phase 1-Cohort 1: GSK2110183 50 mg
Arm/Group | Phase 1 (Dose Escalation)-Cohort 1: GSK2110183 50 mg | Phase 1 (Dose Escalation)-Cohort 1.5: GSK2110183 75 mg | Phase 1 (Dose Escalation)-Cohort 2: GSK2110183 100 mg | Phase 1 (Dose Escalation)-Cohort 3: GSK2110183 125 mg | Phase 1 (Dose Escalation)-Cohort 4: GSK2110183 150 mg | Phase 2 (Treatment Group): GSK2110183 125 mg (MTD)
Started | 4 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1-Cohort 1.5: GSK2110183 75 mg
Arm/Group | Phase 1 (Dose Escalation)-Cohort 1: GSK2110183 50 mg | Phase 1 (Dose Escalation)-Cohort 1.5: GSK2110183 75 mg | Phase 1 (Dose Escalation)-Cohort 2: GSK2110183 100 mg | Phase 1 (Dose Escalation)-Cohort 3: GSK2110183 125 mg | Phase 1 (Dose Escalation)-Cohort 4: GSK2110183 150 mg | Phase 2 (Treatment Group): GSK2110183 125 mg (MTD)
Started | 0 | 4 | 0 | 0 | 0 | 0
Completed | 0 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Clinical Progression | 0 | 1 | 0 | 0 | 0 | 0
Period: Phase 1-Cohort 2: GSK2110183 100 mg
Arm/Group | Phase 1 (Dose Escalation)-Cohort 1: GSK2110183 50 mg | Phase 1 (Dose Escalation)-Cohort 1.5: GSK2110183 75 mg | Phase 1 (Dose Escalation)-Cohort 2: GSK2110183 100 mg | Phase 1 (Dose Escalation)-Cohort 3: GSK2110183 125 mg | Phase 1 (Dose Escalation)-Cohort 4: GSK2110183 150 mg | Phase 2 (Treatment Group): GSK2110183 125 mg (MTD)
Started | 0 | 0 | 6 | 0 | 0 | 0
Completed | 0 | 0 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0
Period: Phase 1-Cohort 3: GSK2110183 125 mg
Arm/Group | Phase 1 (Dose Escalation)-Cohort 1: GSK2110183 50 mg | Phase 1 (Dose Escalation)-Cohort 1.5: GSK2110183 75 mg | Phase 1 (Dose Escalation)-Cohort 2: GSK2110183 100 mg | Phase 1 (Dose Escalation)-Cohort 3: GSK2110183 125 mg | Phase 1 (Dose Escalation)-Cohort 4: GSK2110183 150 mg | Phase 2 (Treatment Group): GSK2110183 125 mg (MTD)
Started | 0 | 0 | 0 | 12 | 0 | 0
Completed | 0 | 0 | 0 | 10 | 0 | 0
Not Completed | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Clinical Progression | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Period: Phase 1-Cohort 4: GSK2110183 150 mg
Arm/Group | Phase 1 (Dose Escalation)-Cohort 1: GSK2110183 50 mg | Phase 1 (Dose Escalation)-Cohort 1.5: GSK2110183 75 mg | Phase 1 (Dose Escalation)-Cohort 2: GSK2110183 100 mg | Phase 1 (Dose Escalation)-Cohort 3: GSK2110183 125 mg | Phase 1 (Dose Escalation)-Cohort 4: GSK2110183 150 mg | Phase 2 (Treatment Group): GSK2110183 125 mg (MTD)
Started | 0 | 0 | 0 | 0 | 3 | 0
Completed | 0 | 0 | 0 | 0 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2: GSK2110183 125 mg
Arm/Group | Phase 1 (Dose Escalation)-Cohort 1: GSK2110183 50 mg | Phase 1 (Dose Escalation)-Cohort 1.5: GSK2110183 75 mg | Phase 1 (Dose Escalation)-Cohort 2: GSK2110183 100 mg | Phase 1 (Dose Escalation)-Cohort 3: GSK2110183 125 mg | Phase 1 (Dose Escalation)-Cohort 4: GSK2110183 150 mg | Phase 2 (Treatment Group): GSK2110183 125 mg (MTD)
Started | 0 | 0 | 0 | 0 | 0 | 30 (Per SAP, Cohort B (n=2) data was summarized in phase 2 total column as cohort B had <10 subjects.)
Completed | 0 | 0 | 0 | 0 | 0 | 22
Not Completed | 0 | 0 | 0 | 0 | 0 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Clinical Progression | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase 1 (Dose Escalation): GSK2110183: GSK2110183, either at 50 mg, 75 mg, 100 mg, 125 mg or 150 mg capsule by mouth daily in combination with carboplatin AUC 5 and paclitaxel 175 mg/m2 given intravenously every 3 weeks for a maximum 6 cycles.
- Phase 2 (Treatment Group): GSK2110183: The dosing regimen identified in Phase 1 will then be evaluated in Phase 2, a single arm study focused on clinical efficacy. GSK2110183 125 mg (MTD) capsule by mouth daily in combination with carboplatin AUC 5 and paclitaxel 175 mg/m2 given intravenously every 3 weeks for a maximum 6 x 21 day cycles followed by continuous GSK2110183 150 mg capsule by mouth daily until progression, death or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Phase 1 (Dose Escalation): GSK2110183 | Phase 2 (Treatment Group): GSK2110183 | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Customized [Number; unit: participants]
  18 - 64 years | 18 | 15 | 33
  65 - 84 years | 11 | 15 | 26
Sex/Gender, Customized [Number; unit: participants]
  Female | 29 | 30 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 30 | 59
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 13 | 15 | 28
  United Kingdom | 16 | 10 | 26
  Russian Federation | 0 | 5 | 5
Height [Mean (Standard Deviation); unit: cm] | 160.81 (6.609) | 160.92 (6.016) | 160.86 (6.264)
Weight [Mean (Standard Deviation); unit: kg] | 68.01 (15.847) | 69.45 (15.836) | 68.74 (15.721)

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Subjects With Treatment-Emergent Adverse Events (TEAE) of Grade Greater Than or Equal to (≥) 3 in Severity
Time Frame: Up to Week 3
Population: All Treated Subjects (ATS) in Phase 1.
Measure: Number; unit: Participants
Arm/Group | Phase 1 (Dose Escalation): GSK2110183
Number analyzed (Participants) | 29
Participants
  Subjects with at Least 1 TEAE of Grade ≥3 | 26
  Neutropenia | 12
  Hypomagnesaemia | 6
  Diarrhoea | 1
  Rash Maculo-Papular | 2
  Vomiting | 2
  Anaemia | 3
  Rash | 2
  Fatigue | 1
  Nausea | 3
  Neutropenic sepsis | 1
  Hyperglycemia | 3

2. Primary Outcome: Phase 1 Safety: Number of Subjects Reporting Adverse Events
Description: Study Treatment refers to GSK2110183 with or without Carboplatin and/or Paclitaxel.
  Dose limiting toxicity (DLT): An event is considered a DLT if it had a reasonable causal relationship to study drug & occurs within first 3 weeks of therapy & met at least one of the following criteria:
  * Grade 3 or 4 non-hematologic toxicity as described in the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v4.0, 2009 [NCI, 2009] with the exceptions of Grade 3 electrolyte disturbances that respond to correction within 24 hours; or Grade 3 rash, diarrhea, nausea, vomiting and mucositis that responded to standard medical supportive care within 48 hours).
  * Grade 4 neutropenia lasting ≥5 days
  * Febrile neutropenia
  * Grade 3 thrombocytopenia with bleeding
  * Grade 4 thrombocytopenia
  * Grade 4 anemia
  * Treatment delay of >14 days due to unresolved toxicity
  * Alanine aminotransferase (ALT) >3 times upper limit of normal (ULN) with bilirubin >2 times ULN
Time Frame: Up to Week 3
Population: ATS population (Phase 1)
Measure: Number; unit: participants
Arm/Group | Phase 1 (Dose Escalation): GSK2110183
Number analyzed (Participants) | 29
participants
  Treatment Emergent Adverse Events (TEAEs) | 29
  Serious TEAEs | 14
  GSK2110183 Related Serious TEAEs | 7
  GSK2110183 Related TEAEs | 29
  Study Treatment Related TEAEs | 29
  TEAEs Leading to Discontinuation of GSK2110183 | 6
  TEAEs Leading to Discontinuation of Study Treatmnt | 17
  TEAEs Leading to Dose Modification of GSK2110183 | 18
  TEAEs Leading to Dose Modification of Study Trtmnt | 26
  TEAEs Leading to Death | 0
  Dose Limiting Toxicity | 3

3. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD) of GSK2110183
Description: MTD is defined as the highest dose at which 1 or fewer of up to 6 subjects experience a dose limiting toxicity (DLT) during the first 3 weeks of combination therapy. MTD was considered exceeded if 2 or more subjects in a cohort of up to 6 subjects experienced a DLT.
Time Frame: Up to Week 3
Population: ATS population (Phase 1).
Measure: Number; unit: mg
Arm/Group | Phase 1 (Dose Escalation): GSK2110183
Number analyzed (Participants) | 29
mg | 125

4. Primary Outcome: Overall Response Rate (ORR) in Phase 2 Subjects With Recurrent Platinum-resistant Ovarian Cancer (Cohort A)
Description: Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST) 1.1 criteria for target lesions and assessed by MRI: Complete Response (CR) is Disappearance of all target lesions and Partial Response (PR) is greater than or equal to (≥) 30% decrease in the sum of the longest diameter of target lesions.
  Overall Response (OR) = CR + PR.
Time Frame: Every 3 weeks up to 6 months
Population: ATS population (Phase 2-Cohort A)
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 2 (Treatment Group): GSK2110183
Number analyzed (Participants) | 28
Percentage of participants
  Complete Response | 7.1
  Partial Response | 25.0
  Stable Disease | 39.3
  Progressive Disease | 14.3
  Not Evaluable | 14.3
  Overall Response Rate | 32.1

5. Primary Outcome: ORR in Phase 2 Subjects With Recurrent Platinum-refractory Ovarian Cancer (Cohort B)
Description: Per RECIST version 1.1 criteria for target lesions and assessed by MRI: Complete Response (CR) is Disappearance of all target lesions and Partial Response (PR) is ≥30% decrease in the sum of the longest diameter of target lesions.
  Overall Response (OR) = CR + PR.
Time Frame: Every 3 weeks up to 6 months
Population: As described in SAP (dated 14-Jul-2015), data was not analyzed separately for Cohort B (n=2) as there were <10 subjects in this group due to difficulty in enrolling Platinum-refractory ovarian cancer subjects.
Arm/Group | Phase 2 (Treatment Group): GSK2110183
Number analyzed (Participants) | 0

6. Secondary Outcome: ORR in Phase 1 Subjects With Recurrent Platinum-resistant Ovarian Cancer
Description: as for outcome 5
Time Frame: Up to Week 3
Population: ATS population (Phase 1)
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 1 (Dose Escalation): GSK2110183
Number analyzed (Participants) | 29
Percentage of participants
  Complete Response | 0
  Partial Response | 24.1
  Stable Disease | 44.8
  Progressive Disease | 20.7
  Not Evaluable | 10.3
  Overall Response Rate | 24.1

7. Secondary Outcome: Phase 2: Number of Subjects With Treatment-Emergent Adverse Events (TEAE) of Grade ≥3 in Severity
Time Frame: Up to Day 21 (Phase 2)
Population: ATS population (Phase 2)
Measure: Number; unit: participants
Arm/Group | Phase 2 (Treatment Group): GSK2110183
Number analyzed (Participants) | 30
participants
  Subjects with at Least 1 TEAE of Grade ≥3 | 26
  Neutropenia | 1
  Hypomagnesaemia | 3
  Diarrhoea | 6
  Rash Maculo-Papular | 5
  Vomiting | 4
  Anaemia | 3
  Rash | 3
  Fatigue | 4
  Nausea | 1
  Neutropenic sepsis | 3
  Hyperglycemia | 0

8. Secondary Outcome: Phase 2 Safety: Number of Subjects Reporting Adverse Events
Description: Dose limiting toxicity (DLT): An event is considered a DLT if it had a reasonable causal relationship to study drug & occurs within first 3 weeks of therapy & met at least one of the following criteria:
  * Grade 3 or 4 non-hematologic toxicity as described in the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v4.0, 2009 [NCI, 2009] with the exceptions of Grade 3 electrolyte disturbances that respond to correction within 24 hours; or Grade 3 rash, diarrhea, nausea, vomiting and mucositis that responded to standard medical supportive care within 48 hours).
  * Grade 4 neutropenia lasting ≥5 days
  * Febrile neutropenia
  * Grade 3 thrombocytopenia with bleeding
  * Grade 4 thrombocytopenia
  * Grade 4 anemia
  * Treatment delay of >14 days due to unresolved toxicity
  * Alanine aminotransferase (ALT) >3 times upper limit of normal (ULN) with bilirubin >2 times ULN
Time Frame: Up to Day 51
Population: ATS population (Phase 2)
Measure: Number; unit: participants
Arm/Group | Phase 2 (Treatment Group): GSK2110183
Number analyzed (Participants) | 30
participants
  TEAEs | 30
  Serious TEAEs | 16
  GSK2110183 Related Serious TEAEs | 11
  GSK2110183 Related TEAEs | 25
  Study Treatment Related TEAEs | 30
  TEAEs Leading to Discontinuation of GSK2110183 | 9
  TEAEs Leading to Discontinuation of Study Treatmnt | 13
  TEAEs Leading to Dose Modification of GSK2110183 | 17
  TEAEs Leading to Dose Modification of Study Trtmnt | 24
  TEAEs Leading to Death | 0
  Dose Limiting Toxicity | 0

9. Secondary Outcome: Phase 2: Response Rate (RR) Defined by Gynecologic Cancer Intergroup (GCIG) CA 125
Description: RR is defined by the percentage of subjects with investigator-assessed Partial Cancer Antigen (CA) 125 Response (PR) or Complete CA 125 Response (CR) at any time during the study by GCIG CA 125. PR is greater than (>) 50% decrease in CA-125 values from baseline and no clinical or radiological evidence of new lesions. CR is decrease in the CA-125 to within the normal limits and less than (<) 40 IU/mL and no clinical or radiological evidence of disease.
Time Frame: From Month 1 to 6
Population: ATS population (Phase 2)
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 2 (Treatment Group): GSK2110183
Number analyzed (Participants) | 30
Percentage of participants
  Complete CA 125 Response | 16.7
  Partial CA 125 Response | 30.0
  Stable Response | 30.0
  CA 125 Progression | 0
  Not Evaluable | 23.3
  Response rate | 46.7

10. Secondary Outcome: Progression Free Survival (PFS) by RECIST or Clinical Symptomatic Progression of Subjects With Recurrent Platinum-resistant Ovarian Cancer (Phase 2-Cohort A)
Description: PFS was defined as the number of months between date of first GSK2110183 treatment and the earliest date of disease progression by RECIST or clinical symptomatic progression or death due to any cause whichever is earlier. Progression is defined using RECIST version 1.1 as at least a 20% increase in the sum of the longest diameter of target lesion in reference to the smallest sum of the longest diameter recorded since the treatment started.
Time Frame: From first dose until disease progression or death (approximately 36 months)
Population: ATS population (Phase 2-Cohort A)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 (Treatment Group): GSK2110183
Number analyzed (Participants) | 28
Months | 6.5 [4.4 to 8.1]

11. Secondary Outcome: PFS by RECIST of Subjects With Recurrent Platinum-resistant Ovarian Cancer (Phase 2-Cohort A)
Description: PFS was defined as the number of months between date of first GSK2110183 treatment and the earliest date of disease progression by RECIST or death due to any cause whichever is earlier. Progression is defined using RECIST version 1.1 as at least a 20% increase in the sum of the longest diameter of target lesion in reference to the smallest sum of the longest diameter recorded since the treatment started.
Time Frame: From first dose until disease progression or death (approximately 36 months)
Population: ATS population ((Phase 2-Cohort A)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 (Treatment Group): GSK2110183
Number analyzed (Participants) | 28
Months | 7.1 [6.3 to 9.0]

ADVERSE EVENTS:
Time Frame: Up to Day 51
Description: Included Serious Adverse Events (SAEs) and Adverse Events (AEs) for ATS population
Arm/Group | Phase 1 (Dose Escalation): GSK2110183 | Phase 2 (Treatment Group): GSK2110183
Serious Adverse Events (participants affected / at risk) | 14/29 | 16/30
Other Adverse Events (participants affected / at risk) | 29/29 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (Dose Escalation): GSK2110183 (N=29) | Phase 2 (Treatment Group): GSK2110183 (N=30)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 7 (9)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (4)
Abdominal Pain (Gastrointestinal disorders) | 2 (3) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (3)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colonic Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip Swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal Pain (General disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutropenic Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Lower Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Escherichia Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0)
Lobar Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Oral Infection (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Tract Infection Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Influenza Like Illness (General disorders) | 1 (1) | 0 (0)
Mucosal Inflammation (General disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (Dose Escalation): GSK2110183 (N=29) | Phase 2 (Treatment Group): GSK2110183 (N=30)
Diarrhoea (Gastrointestinal disorders) | 23 (45) | 18 (38)
Nausea (Gastrointestinal disorders) | 24 (53) | 15 (20)
Vomiting (Gastrointestinal disorders) | 21 (44) | 14 (22)
Constipation (Gastrointestinal disorders) | 12 (20) | 13 (14)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 14 (25) | 6 (11)
Abdominal pain (Gastrointestinal disorders) | 12 (18) | 6 (8)
Stomatitis (Gastrointestinal disorders) | 8 (14) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 4 (6) | 7 (10)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 3 (3)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 6 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 16 (17) | 16 (17)
Rash (Skin and subcutaneous tissue disorders) | 12 (18) | 5 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 10 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 11 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2)
Fatigue (General disorders) | 19 (37) | 18 (27)
Oedema peripheral (General disorders) | 5 (6) | 2 (4)
Mucosal inflammation (General disorders) | 5 (6) | 1 (1)
Chest pain (General disorders) | 3 (5) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 16 (27) | 14 (22)
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 (10) | 8 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 6 (6) | 6 (6)
Headache (Nervous system disorders) | 8 (11) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (11) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 5 (9)
Neurotoxicity (Nervous system disorders) | 3 (4) | 2 (4)
Dizziness (Nervous system disorders) | 2 (2) | 2 (6)
Paraesthesia (Nervous system disorders) | 0 (0) | 3 (3)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (21) | 7 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (13) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 14 (19) | 5 (6)
Anaemia (Blood and lymphatic system disorders) | 3 (5) | 9 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (7) | 8 (11)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (2) | 3 (4)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (16) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 4 (5)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2) | 1 (2)
Weight decreased (Investigations) | 2 (2) | 1 (1)
White blood cell count decreased (Investigations) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (6) | 6 (6)
Hypertension (Vascular disorders) | 1 (1) | 4 (4)
Hot flush (Vascular disorders) | 1 (1) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 4 (7) | 1 (2)
Hypersensitivity (Immune system disorders) | 1 (2) | 4 (5)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (7) | 1 (1)
CARDIAC DISORDERS (Cardiac disorders) | 2 (2) | 3 (3)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 3 (3) | 2 (9)
EYE DISORDERS (Eye disorders) | 2 (3) | 2 (2)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS (Reproductive system and breast disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No